CLINICAL TRIAL: NCT01192100
Title: The Beneficial Effects of a Protein-rich Breakfast on Appetite Control & Cognition in Overweight and Obese Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: American Egg Board (Other); National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Responsible Party: Principal Investigator, Heather Leidy, Assistant Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1173258
Record Dates: First submitted 2010-08-27; First posted 2010-08-31 (Estimated); Results first posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Overweight; Obesity
Keywords: Protein-rich breakfast; Breakfast Skipping; Adolescents; Obesity; Increased dietary protein; Breakfast; fMRI; Ghrelin; PYY
MeSH Terms: conditions — Overweight; Obesity; Intermittent Fasting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Breakfast Skipping (Experimental): Breakfast skipping serves as the baseline/control arm since the participants habitually skip breakfast (i.e., skip breakfast at least 5 times/week). Thus, during the week prior to and including the testing day, the participants will continue to skip breakfast each morning.
  Interventions: Behavioral: Breakfast Skipping
- Normal Protein Breakfast Meals (Experimental): For 7 days, the participants will consume normal protein breakfast meals each morning. These meals will consist of cereal-based foods and will be 350 kcal, which is approximately 18% of daily energy intake for overweight and obese adolescents ages 9-18 y. The macronutrient composition of these meals will contain 15% protein (13 g of dietary protein), 65% CHO, and 20% fat.
  Interventions: Behavioral: Normal Protein Breakfast Meals
- Protein-rich Breakfast Meals (Experimental): For 7 days, the participants will consume protein-rich breakfast meals each morning. These meals will consist of home-cooked foods and will be 350 kcal, which is approximately 18% of daily energy intake for overweight and obese adolescents ages 9-18 y. The macronutrient composition of these meals will contain 40% protein (35 g of protein), 40% CHO, and 20% fat.
  Interventions: Behavioral: Protein-rich Breakfast Meals

INTERVENTIONS:
Behavioral: Breakfast Skipping — Participants will continue to skip breakfast each morning.
  Other Names: Control
  Arms: Breakfast Skipping
Behavioral: Normal Protein Breakfast Meals — Participants will consume normal protein breakfast meals each morning.
  Arms: Normal Protein Breakfast Meals
Behavioral: Protein-rich Breakfast Meals — Participants will consume protein-rich breakfast meals each morning.
  Arms: Protein-rich Breakfast Meals

SUMMARY:
The purpose of this study is to assess whether the daily addition of a protein-rich breakfast leads to beneficial changes in appetite control, food intake regulation,and cognitive function in overweight & obese 'breakfast skipping' young women.

DETAILED DESCRIPTION:
Breakfast skipping, which is a common, yet unhealthy dietary habit among young women, has been strongly associated with over-eating (especially in the evening), weight gain, and obesity. Breakfast skipping has also been shown to reduce cognitive function in this population. However, it is unclear as to whether the addition of breakfast, with specific emphasis on increased dietary protein, leads to improvements in these outcomes. This study will provide mechanistic evidence supporting the addition of a protein-rich breakfast to improve and/or re-establish appetite control, energy intake regulation, and cognitive function in overweight/obese 'breakfast skipping' young women. 22 overweight and obese 'breakfast skipping' adolescent girls will participate in the following randomized within-subject crossover-design breakfast study. The participants will randomly complete the follow breakfast patterns at home for 6 days: 1) Breakfast Skipping; 2) Consumption of Normal Protein breakfast meals(i.e., 350 kcal; 15% of the meal as protein, 65% CHO, & 20% fat); and 3) Consumption of Protein-Rich breakfast meals (i.e., 350 kcal; 40% of the meal as protein, 40% CHO, & 20% fat). On the 7th day of each pattern, the participants will report to the MU-Brain Imaging Center in the morning to complete the respective 10-h testing day. The participants will begin the testing day by either skipping breakfast or consuming their respective breakfast meal. Blood samples and assessments of perceived appetite, pleasure/reward, and cognitive function will be collected/completed at specific times throughout the day. A standardized lunch will also be provided. Prior to dinner, a brain scan will be completed using functional magnetic resonance imaging (fMRI) to identify brain activation patterns in response to food pictures. Following the fMRI, the participants will be provided with an ad libitum dinner buffet to consume of the facility. They will also be given evening snacks to consume ad libitum, at home throughout the remainder of the day. There is a 7-day washout period between each breakfast pattern. Primary outcomes include morning, mid-day, afternoon, and evening appetite, satiety, pleasure/reward, hormonal responses (plasma glucose, insulin, ghrelin, and PYY concentrations), brain activation patterns, evening energy intake, and daily energy intake.

ELIGIBILITY:
Inclusion Criteria:

The participants must meet the following inclusion criteria:

* Female
* Age range 15-20 y
* Overweight to obese (85th -99th percentile for BMI for age; BMI: 25-39.9 kg/m2
* No metabolic, psychological, or neurological diseases/conditions
* Not currently/previously on a weight loss/other special diet
* Frequently eats lunch ( ≥ 5 eating occasions/wk)
* Consistently skips breakfast every week day (i.e., 5 week days/week)
* Right-handed (necessary for the fMRI analyses)

Exclusion Criteria:

The participants will be excluded from participation in the study if they meet the following exclusion criteria:

* Male
* Age >20 y and <15 y
* Under Weight (<5th percentile for BMI for age; BMI: <18 kg/m2)
* Normal Weight (6th-84th percentile for BMI for age; BMI: 18-24.0 kg/m2)
* Morbidly Obese (BMI: >40 kg/m2)
* Clinically diagnosed with diabetes (Type I or Type II), having an eating disorder, or having any other metabolic, psychological, or neurological diseases/conditions that would influence the study outcomes.
* Not currently/previously on a weight loss or other special diet (in the past 6 months)
* Skip lunch ( ≥ 2 eating occasions/wk)
* Consume breakfast (≥ 2 eating occasions/wk)
* Left-handed
* Claustrophobic (≥ 2 past bouts of claustrophobia when exposure to small spaces)
* Do not meet the fMRI criteria established by the MU-BIC (regarding metal implants, etc.)
* Pregnant

Ages: 15 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Leidy, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leidy HJ, Ortinau LC, Douglas SM, Hoertel HA. Beneficial effects of a higher-protein breakfast on the appetitive, hormonal, and neural signals controlling energy intake regulation in overweight/obese, "breakfast-skipping," late-adolescent girls. Am J Clin Nutr. 2013 Apr;97(4):677-88. doi: 10.3945/ajcn.112.053116. Epub 2013 Feb 27. PMID 23446906

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Protein > High Protein > Skip: 6 overweight 'breakfast skipping' adolescent girls participated in a randomized crossover-design breakfast study where they were completed, in the following order, the follow breakfast patterns at home for 6 days: 1) Consumption of Normal Protein breakfast meals (i.e., 350 kcal; 15% protein, 65% CHO, & 20% fat); 2) Consumption of Protein-Rich breakfast meals (i.e., 350 kcal; 40% protein, 40% CHO, & 20% fat); and 3) Breakfast Skipping. On the 7th day of each pattern, the participants reported to the testing facilities in the morning to complete the respective 10-h testing day. Blood samples and assessments of perceived appetite were collected/completed throughout the day following the breakfast (or no breakfast). A standardized lunch was also be provided. Prior to dinner, a brain scan was completed using functional magnetic resonance imaging (fMRI) to identify brain activation patterns in response to food pictures. There was a 7-day washout period between each breakfast pattern.
- Skip > Normal Protein > High Protein: 4 overweight 'breakfast skipping' adolescent girls participated in a randomized crossover-design breakfast study where they were completed, in the following order, the follow breakfast patterns at home for 6 days: 1) Breakfast Skipping; 2) Consumption of Normal Protein breakfast meals (i.e., 350 kcal; 15% protein, 65% CHO, & 20% fat) and 3) Consumption of Protein-Rich breakfast meals (i.e., 350 kcal; 40% protein, 40% CHO, & 20% fat). On the 7th day of each pattern, the participants reported to the testing facilities in the morning to complete the respective 10-h testing day. Blood samples and assessments of perceived appetite were collected/completed throughout the day following the breakfast (or no breakfast). A standardized lunch was also be provided. Prior to dinner, a brain scan was completed using functional magnetic resonance imaging (fMRI) to identify brain activation patterns in response to food pictures. There was a 7-day washout period between each breakfast pattern.
- Skip > High Protein > Normal Protein: 3 overweight 'breakfast skipping' adolescent girls participated in a randomized crossover-design breakfast study where they were completed, in the following order, the follow breakfast patterns at home for 6 days: 1) Breakfast Skipping; 2) Consumption of Protein-Rich breakfast meals (i.e., 350 kcal; 40% protein, 40% CHO, & 20% fat), and 3) Consumption of Normal Protein breakfast meals (i.e., 350 kcal; 15% protein, 65% CHO, & 20% fat). On the 7th day of each pattern, the participants reported to the testing facilities in the morning to complete the respective 10-h testing day. Blood samples and assessments of perceived appetite were collected/completed throughout the day following the breakfast (or no breakfast). A standardized lunch was also be provided. Prior to dinner, a brain scan was completed using functional magnetic resonance imaging (fMRI) to identify brain activation patterns in response to food pictures. There was a 7-day washout period between each breakfast pattern.
- High Protein > Skip > Normal Protein: 4 overweight 'breakfast skipping' adolescent girls participated in a randomized crossover-design breakfast study where they were completed, in the following order, the follow breakfast patterns at home for 6 days: 1) Consumption of Protein-Rich breakfast meals (i.e., 350 kcal; 40% protein, 40% CHO, & 20% fat), 2) Breakfast Skipping and 3) Consumption of Normal Protein breakfast meals (i.e., 350 kcal; 15% protein, 65% CHO, & 20% fat). On the 7th day of each pattern, the participants reported to the testing facilities in the morning to complete the respective 10-h testing day. Blood samples and assessments of perceived appetite were collected/completed throughout the day following the breakfast (or no breakfast). A standardized lunch was also be provided. Prior to dinner, a brain scan was completed using functional magnetic resonance imaging (fMRI) to identify brain activation patterns in response to food pictures. There was a 7-day washout period between each breakfast pattern
- High Protein > Normal Protein > Skip: 3 overweight 'breakfast skipping' adolescent girls participated in a randomized crossover-design breakfast study where they were completed, in the following order, the follow breakfast patterns at home for 6 days: 1) Consumption of Protein-Rich breakfast meals (i.e., 350 kcal; 40% protein, 40% CHO, & 20% fat), 2) Consumption of Normal Protein breakfast meals (i.e., 350 kcal; 15% protein, 65% CHO, & 20% fat) and 3) Breakfast Skipping. On the 7th day of each pattern, the participants reported to the testing facilities in the morning to complete the respective 10-h testing day. Blood samples and assessments of perceived appetite were collected/completed throughout the day following the breakfast (or no breakfast). A standardized lunch was also be provided. Prior to dinner, a brain scan was completed using functional magnetic resonance imaging (fMRI) to identify brain activation patterns in response to food pictures. There was a 7-day washout period between each breakfast pattern.
- Normal Protein > Skip > High Protein: 2 overweight 'breakfast skipping' adolescent girls participated in a randomized crossover-design breakfast study where they were completed, in the following order, the follow breakfast patterns at home for 6 days: 1) Consumption of Normal Protein breakfast meals (i.e., 350 kcal; 15% protein, 65% CHO, & 20% fat), 2) Breakfast Skipping and 3) Consumption of Protein-Rich breakfast meals (i.e., 350 kcal; 40% protein, 40% CHO, & 20% fat). On the 7th day of each pattern, the participants reported to the testing facilities in the morning to complete the respective 10-h testing day. Blood samples and assessments of perceived appetite were collected/completed throughout the day following the breakfast (or no breakfast). A standardized lunch was also be provided. Prior to dinner, a brain scan was completed using functional magnetic resonance imaging (fMRI) to identify brain activation patterns in response to food pictures. There was a 7-day washout period between each breakfast pattern.
Period: Overall Study
Arm/Group | Normal Protein > High Protein > Skip | Skip > Normal Protein > High Protein | Skip > High Protein > Normal Protein | High Protein > Skip > Normal Protein | High Protein > Normal Protein > Skip | Normal Protein > Skip > High Protein
Started | 6 | 4 | 3 | 4 | 3 | 2
Began 1st Intervention Week | 6 | 4 | 3 | 4 | 3 | 2
Began 2nd Intervention Week | 6 | 4 | 3 | 3 | 2 | 2
Began 3rd Intervention Week | 6 | 4 | 3 | 3 | 2 | 2
Completed | 6 | 4 | 3 | 3 | 2 | 2
Not Completed | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: 22 overweight 'breakfast skipping' adolescent girls participated in a randomized crossover-design breakfast study where they were completed, in a random order, the follow breakfast patterns at home for 6 days: 1) Breakfast Skipping; 2) Consumption of Normal Protein breakfast meals (i.e., 350 kcal; 15% protein, 65% CHO, & 20% fat); and 3) Consumption of Protein-Rich breakfast meals (i.e., 350 kcal; 40% protein, 40% CHO, & 20% fat). On the 7th day of each pattern, the participants reported to the testing facilities in the morning to complete the respective 10-h testing day. Blood samples and assessments of perceived appetite were collected/completed throughout the day following the breakfast (or no breakfast). A standardized lunch was also be provided. Prior to dinner, a brain scan was completed using functional magnetic resonance imaging (fMRI) to identify brain activation patterns in response to food pictures. There was a 7-day washout period between each breakfast pattern.
Arm/Group | All Study Participants
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 19 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (niAUC) of Perceived Hunger, Fullness, Desire to Eat, and Prospective Food Consumption
Description: Computerized questionnaires, assessing perceived sensations of hunger and fullness were completed throughout the testing days beginning at baseline and about every 30 minutes for a total of 20 questionnaires (- 15 min, +0 min,+30 min, +60 min, +90 min, +120 min, +150 min, +180 min, +210 min, +240 min, +255 min, +270 min, +285 min, +300 min, +330 min, +360 min, +390 min, +420 min, +450 min, and +480 min). The questions are worded as "how strong is your feeling of" with anchors of "not at all" to "extremely." Each reported score can be a minimum of 0 and a maximum of 100 mm. niAUC was calculated by computing the summation of the average change from baseline score (mm) for each time point and the subsequent time point, multiplied by the difference in time (min) between the two measures. For reported feelings of hunger, a higher score can be interpreted as "feeling more hungry" throughout the day. This can be applied to the three other perceived sensations.
Time Frame: 5 weeks
Measure: Mean (Standard Error); unit: mm*min
Arm/Group | Breakfast Skipping | Normal Protein Breakfast Meals | Protein-rich Breakfast Meals
Number analyzed (Participants) | 20 | 20 | 20
mm*min
  How strong is your feeling of hunger? | 17000 (5000) | 11000 (3000) | 10000 (3000)
  How strong is your feeling of being full? | 21000 (5000) | 27000 (6000) | 28000 (8000)
  How strong is your desire to eat? | 18000 (5000) | 13000 (4000) | 12000 (4000)
  How much food can you eat right now? | 17000 (6000) | 13000 (4000) | 10000 (3000)

2. Primary Outcome: Area Under the Curve (AUC) of Plasma Total Ghrelin and Ln Peptide YY (PYY)
Description: The samples were collected in test tubes containing ethylenediaminetetraacetic acid. Protease inhibitors (pefabloc SC and dipeptidyl peptidase) were added to some of the tubes to reduce protein degradation. The plasma was separated and stored in microcentrifuge tubes at -80°C for future analysis. Plasma total ghrelin and peptide YY (PYY) were measured for all time points using the Milliplex multi-analyte profiling magnetic bead-based multi-analyte, metabolic panel, 2-plex assay and Magpix Luminex technologies. AUC was calculated by computing the summation of the average change from baseline score (pg/ml) for each time point and the subsequent time point multiplied by the difference in time (min) between the two time instances for a total of 20 blood samples (- 15 min, +0 min,+30 min, +60 min, +90 min, +120 min, +150 min, +180 min, +210 min, +240 min, +255 min, +270 min, +285 min, +300 min, +330 min, +360 min, +390 min, +420 min, +450 min, and +480 min).
Time Frame: 5 weeks
Measure: Mean (Standard Error); unit: (pg*min)/ml
Arm/Group | Breakfast Skipping | Normal Protein Breakfast Meals | Protein-rich Breakfast Meals
Number analyzed (Participants) | 20 | 20 | 20
(pg*min)/ml
  Ghrelin (10^3) | 41 (4) | 35 (3) | 34 (3)
  Ln PYY | 0 (25) | 90 (80) | 160 (70)

3. Primary Outcome: Brain Regions Displaying Differential Activation Prior to Dinner in Response to Food vs Nonfood Stimuli From Food Cue-stimulate fMRI Brain Scans
Description: Participants viewed 3 categories of pictures including food, nonfood (animals), and blurred baseline images. The pictures from each category were presented in blocks of images. Animal pictures were used to control for visual richness and general interest (i.e., appealing but not appetizing). To determine the effects of breakfast/no breakfast on neural activity associated with food motivation, repeated measures ANOVAs were performed on the brain activation maps within the Brain Voyager software with use of stimulus [food (i.e., appetizing and appealing) vs. nonfood (i.e., animal, nonappetizing but appealing]. To identify significant activations in a priori regions, a cluster level statistical threshold was applied to correct for multiple comparisons. By using this approach, significance was set at P = 0.01, with a cluster-level false-positive rate of a = 0.05
Time Frame: 5 weeks
Population: Coordinates were only determined for regions considered significant by analysis using Brain Voyager.
Measure: Number; unit: Talairach Coordinates
Groups:
- Activation After Skipping Breakfast is > After Consuming: To determine the effects of breakfast/no breakfast on neural activity associated with food motivation, repeated measures ANOVAs were performed on the brain activation maps within the Brain Voyager software with use of stimulus [food (i.e., appetizing and appealing) vs. nonfood (i.e., animal, nonappetizing but appealing]. Talairach coordinates for each region are presented for each row as (x;y;z) when activation was determined significant.
- Activation After Normal-protein Breakfast is > After High: For 7 days, the participants will consume normal protein breakfast meals each morning. These meals will consist of cereal-based foods and will be 350 kcal, which is approximately 18% of daily energy intake for overweight and obese adolescents ages 9-18 y. The macronutrient composition of these meals will contain 15% protein (13 g of dietary protein), 65% CHO, and 20% fat.
  Normal Protein Breakfast Meals: Participants will consume normal protein breakfast meals each morning.
Arm/Group | Activation After Skipping Breakfast is > After Consuming | Activation After Normal-protein Breakfast is > After High
Number analyzed (Participants) | 20 | 20
Talairach Coordinates
  Amygdala (x): number analyzed (Participants) | 20 | 0
  Amygdala (x) | -28 |
  Amygdala (y): number analyzed (Participants) | 20 | 0
  Amygdala (y) | -5 |
  Amygdala (z): number analyzed (Participants) | 20 | 0
  Amygdala (z) | -18 |
  Hippocampus (x) | -31 | -19
  Hippocampus (y) | -11 | -17
  Hippocampus (z) | -12 | -18
  Middle Frontal Gyrus (x): number analyzed (Participants) | 20 | 0
  Middle Frontal Gyrus (x) | -25 |
  Middle Frontal Gyrus (y): number analyzed (Participants) | 20 | 0
  Middle Frontal Gyrus (y) | -8 |
  Middle Frontal Gyrus (z): number analyzed (Participants) | 20 | 0
  Middle Frontal Gyrus (z) | 42 |
  Parahippocampus (x): number analyzed (Participants) | 0 | 20
  Parahippocampus (x) |  | -28
  Parahippocampus (y): number analyzed (Participants) | 0 | 20
  Parahippocampus (y) |  | -17
  Parahippocampus (z): number analyzed (Participants) | 0 | 20
  Parahippocampus (z) |  | -30

4. Secondary Outcome: Daily Energy Intake
Description: Energy intake during breakfast, lunch, dinner, and evening snacks of each testing day will be measured.
Time Frame: 5 weeks
Measure: Mean (Standard Error); unit: kilocalories
Arm/Group | Breakfast Skipping | Normal Protein Breakfast Meals | Protein-rich Breakfast Meals
Number analyzed (Participants) | 20 | 20 | 20
kilocalories | 2002 (111) | 2292 (115) | 2123 (71)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Breakfast Skipping | Normal Protein Breakfast Meals | Protein-rich Breakfast Meals
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No